CLINICAL TRIAL: NCT04452097
Title: A Phase 1/2a Study of the Safety and Efficacy of BX-U001 for the Treatment of Severe COVID-19 Pneumonia With Moderate to Severe Acute Respiratory Distress Syndrome (ARDS).
Brief Title: Use of hUC-MSC Product (BX-U001) for the Treatment of COVID-19 With ARDS
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It is a strategic decision by the company, coupled with low incidence of ARDS cases following widespread vaccination efforts.
Sponsor: Baylx Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BXU001-COVID19
Record Dates: First submitted 2020-06-28; First posted 2020-06-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; ARDS; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: In phase 1, eligible subjects will be divided into low, medium and high-dose groups with 3 patients/group. If there is no safety concerns for each group, the dose will be escalated from lower dose to the next higher dose. In phase 2a, a total of 30 subjects will be randomized into the treatment and control groups with a ratio of 3:2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase 1 Low-dose Group (Experimental): Eligible subjects will receive a single infusion of hUC-MCS product at the dose of 0.5 million cells/kg in addition to standard of care treatment.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells + best supportive care
- Phase 1 Middle-dose Group (Experimental): Eligible subjects will receive a single infusion of hUC-MCS product at the dose of 1 million cells/kg in addition to standard of care treatment.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells + best supportive care
- Phase 1 High-dose Group (Experimental): Eligible subjects will receive a single infusion of hUC-MCS product at the dose of 1.5 million cells/kg in addition to standard of care treatment.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells + best supportive care
- Phase 2a Treatment Group (Experimental): Eligible subjects will receive a single infusion of hUC-MCS product at the selected dose from phase 1 in addition to standard of care treatment.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells + best supportive care
- Phase 2a Control Group (Placebo Comparator): Eligible subjects will receive a single infusion of placebo control and standard of care treatment.
  Interventions: Other: Placebo control + best supportive care

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells + best supportive care — hUC-MSC product will be administered intravenously in addition to the standard of care treatment.
  Arms: Phase 1 High-dose Group; Phase 1 Low-dose Group; Phase 1 Middle-dose Group; Phase 2a Treatment Group
Other: Placebo control + best supportive care — Placebo control will be administered intravenously in addition to the standard of care treatment.
  Arms: Phase 2a Control Group

SUMMARY:
This is a phase 1/2a study including 2 parts, phase 1 and phase 2a. The phase 1 part is an open-label, single-arm, dose-escalating study to evaluate the safety and explore the dose limiting toxicity and maximum tolerated dose of a human umbilical cord derived mesenchymal stem cell product (BX-U001) in severe COVID-19 pneumonia patients with acute respiratory distress syndrome (ARDS). Qualified subjects after the screening will be divided into low, medium, or high dose groups to receive a single intravenous infusion of BX-U001 at the dose of 0.5×10^6, 1.0×10^6, or 1.5×10^6 cells/kg of body weight, respectively. The Phase 2a part is a randomized, placebo-controlled, double-blind clinical trial examining the safety and biological effects of BX-U001 at the appropriate dose selected from phase 1 for severe COVID-19 pneumonia patients with the same inclusion/exclusion criteria as the phase 1 part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged between 18 and 80;
2. Laboratory (RT-PCR, Gene Sequencing or Antibody) confirmed cases of severe COVID-19 pneumonia with mild to moderate ARDS (Berlin definition);
3. Patients are intubated;
4. Patients who voluntarily adhere to the research procedures and ensure good compliance during the research period;
5. Patients who fully understand the research nature of this study and sign written informed consent.

Exclusion Criteria:

1. Subjects who have received investigational drug (except for Remdesivir) for the treatment of COVID-19 within 30 days before screening;
2. Subjects who are pregnant, breastfeeding or whose urinary pregnancy test is positive before participation in the study; subjects who are pregnant, breastfeeding, have a birth plan, or are unwillingness to use contraception during the study period and within 12 months of infusion; except for subjects who have sterilization surgery or menopause during the study period;
3. Within 3 days before screening/randomization, subjects who have used high-dose corticosteroids that is equivalent to methylprednisolone >240 mg/day or irregular use of systemic corticosteroids to treat other diseases that could affect the efficacy evaluated by the investigator;
4. Subjects receiving extracorporeal membrane oxygenation (ECMO) support.
5. Subjects who are allergic to low-molecular-weight heparin calcium or human albumin;
6. Subjects with ongoing malignant tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of infusion-related adverse events | Day 3
  Safety will be defined by the incidence of infusion-related adverse events as assessed by the treating physician
Incidence of any treatment-emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) | Day 28
  Safety will be defined by the incidence of TEAEs and TESAEs as assessed by the treating physician

SECONDARY OUTCOMES:
Selection of an appropriate dose of BX-U001 for the following Phase 2 study | Day 28
  The dose will be selected based on the assessment of dose-limiting toxicity and maximum tolerated dose.
All-cause mortality | Day 28
Proportion of patients achieving clinical response by the improvement of at least 2 points on the 7-point ordinal scale. | Day 14
  The scale is as follows: 1. Death 2. Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO) 3. Hospitalized, on non-invasive ventilation or high flow oxygen devices 4. Hospitalized, requiring low flow supplemental oxygen 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise) 6. Hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care 7. Not hospitalized.
Duration of ICU stay | Day 28
Duration of hospital stay | Day 28
Changes in blood cytokine levels | Day 28